CLINICAL TRIAL: NCT01535482
Title: Cognitive Therapy for Suicidal Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH086572-01A2 (NIH); 1R01MH086572-01A2 (NIH)
Record Dates: First submitted 2011-08-25; First posted 2012-02-17 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Suicide, Attempted
Keywords: Cognitive therapy; Suicide; Older men; suicide ideation
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Therapy (Experimental): A cognitive therapy protocol specifically designed to target suicidal ideation in older adults.
  Interventions: Behavioral: Cognitive Therapy
- Enhanced Usual Care (Active Comparator): Enhanced usual care consists of the usual care that individuals receive for suicide prevention, plus assessment and referral services provided by project staff, and weekly phone calls provided by study therapists.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Cognitive Therapy — Cognitive therapy (CT) will consist of 12 to 16 individual CT sessions on a weekly basis plus 3 booster sessions.
  Arms: Cognitive Therapy
Behavioral: Enhanced Usual Care — Enhanced usual care (EUC) will consist of the usual care that individuals receive for suicide prevention in the community, assessment and referral services provided by study staff, and weekly telephone calls lasting 15-30 minutes provided by study therapists to ensure patient safety and to provide some support.
  Arms: Enhanced Usual Care

SUMMARY:
The primary aim of the proposed study is to compare the efficacy of cognitive therapy (CT) with the efficacy of an enhanced usual care (EUC) intervention for reducing the rate of suicide ideation (SI) and the severity of depression and hopelessness among older men. The investigators expect that suicidal older men randomly assigned to the CT intervention condition will have a lower rate of SI during the follow-up period than participants assigned to the control condition.

DETAILED DESCRIPTION:
Older adult males have the highest suicide rate of any age group in the U.S. However, most research concerning treatments for suicide ideation and behavior has focused on adolescents and young adults. Very few treatments have been developed to reduce suicide ideation and behavior in men aged 50 and above. This study will assess the effectiveness of specialized cognitive therapy versus enhanced usual care in treating older men with suicide ideation.

Participants in this five-year study will be randomly assigned to receive either cognitive therapy or enhanced usual care. Participants will be identified within the VA Medical Center and the University of Pennsylvania Health System (UPHS) as having experienced suicide ideation in the past month. Cognitive therapy will be provided by Ph.D.-level therapists and will be geared specifically toward older men with suicidal tendencies. The enhanced usual care condition will consist of the usual care that individuals receive for suicide prevention, plus assessment and referral services provided by independent evaluators and study case managers. In addition, patients in the enhanced usual care condition will receive weekly telephone calls from the study therapists. These phone calls will be approximately 15-30 minutes in duration and their purpose will be to ensure patient safety and to provide some support. All participants will be assessed pre-treatment to attain baseline measures of suicide ideation, hopelessness, and depression. Study visits will occur at baseline and Months 1, 3, 6, 9, and 12 to assess suicide ideation. Self-report and clinician-administered measures will be used to assess participants' progress.

ELIGIBILITY:
Inclusion Criteria:

1. Suicidal intent or desire during the past month prior to the baseline interview as indicated by a score of 1 or higher on items 4 or 5 of the Scale for Suicide Ideation.
2. Male
3. 50 years of age or older
4. Able to speak English
5. Able to provide written informed consent
6. Able to attend study assessment and therapy sessions
7. Able to provide at least two verifiable contacts for tracking purposes
8. Able to function at an intellectual level to allow for the reliable completion of study assessments and participate in psychotherapy as indicated by a Mini-Mental Status Exam (MMSE) total score of 24 or higher and an Executive Interview (EXIT-25) total score of 14 or lower.

Exclusion Criteria:

1. Needed priority treatment for a substance use disorder as determined by the referring clinician.
2. Needed priority treatment for PTSD as determined by the referring clinician.
3. Taking antidepressant medication for less than one month, or if antidepressant medication has been changed in the last month as indicated by the Alexopolous "Composite Antidepressant Score" Scale.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Change in baseline suicidal ideation | baseline, 1, 3, 6, 9, 12 months

SECONDARY OUTCOMES:
depression | baseline, 1, 3, 6, 9, 12 months
hopelessness | baseline, 1, 3, 6, 9, 12 months
quality of life | baseline, 1, 3, 6, 9, 12 months
social problem solving skills | baseline, 1, 3, 6, 9, 12 months
complicated grief | baseline, 1, 3, 6, 9, 12 months
reasons for living and dying | baseline, 1, 3, 6, 9, 12 months
perceived social support | baseline, 1, 3, 6, 9, 12 months
Cognitive Executive Functioning | baseline, 1, 3, 6, 9, 12 months
  Executive functioning will be measured by scores on an Executive Functioning Interview, which measures skills such as planning, working memory, attention, inhibition, and mental flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Aaron T. Beck Psychopathology Research Center - University of Pennsylvania, Philadelphia, Pennsylvania, United States